CLINICAL TRIAL: NCT06728579
Title: Enhanced Pain Coping in Cancer (EPIC): A Study of Managing Treatment-Related Joint Pain in Breast Cancer Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-171
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Survivor
Keywords: Enhanced Pain Coping in Cancer; Mindfulness Oriented Recovery Enhancement; Aromatase inhibitors; Arthralgia; Ache; Cancer Pain; Cancer Survivors
MeSH Terms: conditions — Arthralgia; Pain; Cancer Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel group, RCT
Who Masked: Investigator, Outcomes Assessor
Masking Description: This is a double-blind study where PIs, biostatisticians, and the CRC who performs outcome assessments are blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MORE Treatment Group (Experimental): Participants randomized to the MORE arm will participate in eight weekly, two-hour group sessions following an established protocol. MORE sessions involve instruction in three therapeutic skills: 1) mindfulness to reduce pain and increase self regulation over maladaptive pain coping habits, (2) reappraisal to decrease psychological distress and negative affect, and 3) savoring to amplify natural reward processing and evoke positive emotion (see Figure 2). Participants will be asked to engage in 15 minutes per day of skill practice at home guided by audio recording, and to record the number of minutes they engaged in skill practice via a weekly Research Electronic Data Capture (REDCap) survey.
  Interventions: Behavioral: Mindfulness Oriented Recovery Enhancement (MORE); Other: Questionnaires
- Supportive Psychotherapy Control Group (Active Comparator): Participants randomized to SG will participate in eight weekly two-hour SG sessions led by the same instructors who deliver MORE interventions. The instructors will lead discussions on themes pertinent to chronic pain and cancer survivorship (see Figure 3) but will not teach MORE skills. To match the MORE homework requirement, SG participants will be asked to journal for 15 minutes/day on weekly session topics. Providers will employ empathic responding, elicit emotional expression, and promote a positive group climate.
  Interventions: Other: Questionnaires; Behavioral: Supportive Psychotherapy (SG)

INTERVENTIONS:
Behavioral: Mindfulness Oriented Recovery Enhancement (MORE) — eight weekly two-hour MORE sessions
  Arms: MORE Treatment Group
Other: Questionnaires — filled out up to 24 weeks
Behavioral: Supportive Psychotherapy (SG) — eight weekly two-hour SG sessions
  Arms: Supportive Psychotherapy Control Group

SUMMARY:
The researchers are doing this study to compare two different types of group therapy and find out whether they are effective approaches for helping breast cancer survivors manage joint pain caused by aromatase inhibitors (AI). This type of joint pain is called AI-associated arthralgia, or AIA, and it is common in people taking AIs. AIA and its associated symptoms can make some people decide to stop taking their medication. The study will look at the effects of two different types of group therapy on participants' cancer-related symptoms (such as pain, fatigue, and anxiety), their ability to continue taking AIs on a regular schedule, and their quality of life. We will measure participants' quality of life by having them fill out questionnaires.

Both groups will have 2-hour group therapy sessions once a week, over the course of 8 weeks. During the sessions, you will be in a group of 6-10 participants, who may be a mixture of patients from both MSK and University of California San Diego (UCSD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* English-proficient women with a history of stage I, II, or III breast cancer
* Free of oncologic disease by clinical examination and history;
* Receiving third-generation AI therapy (anastrozole, letrozole, or exemestane) for at least 28 days prior to consent with plan to continue for at least another 12 months;
* Worst joint pain rated at least 4 or greater on a 0-10 numeric rating scale in the preceding week prior to consent;
* Reporting at least 15 days with pain in the preceding 30 days prior to consent;
* Experiencing joint pain for at least one month;
* Pain attributed to AI therapy;
* Willing to adhere to all study-related procedures, including randomization to one of two treatment arms: Mindfulness-Oriented Recovery Enhancement (MORE) or Supportive Group Psychotherapy (SG);
* Able to attend video-call sessions in a quiet/private location.

Exclusion Criteria:

* Metastatic breast cancer (stage IV);
* Completed chemotherapy, surgery, or radiation therapy less than 4 weeks prior to enrollment;
* Pain attributed to inflammatory arthritis (i.e. rheumatoid arthritis, gout, pseudogout);
* Surgery or joint injection involving the affected joints within the last month or planned within the next six months;
* Active suicidality or psychosis as determined by the Mini-International Neuropsychiatric Interview.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 200 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pain Interference | up to 24 weeks
  Pain interference will be assessed using the 7-item Pain Interference subscale from the Brief Pain Inventory Short Form (BPI-SF). Each item is rated on a scale from 0 ("does not interfere") to 10 ("completely interferes"), with higher scores indicating worse interference. The BPI is a widely used, reliable, valid, and responsive tool for measuring pain (Cronbach's α 0.77-0.91). The Pain Interference subscale will be administered at baseline, weekly during the 8-week intervention, and at weeks 12 and 24. Completing the survey requires approximately 1 minute.

SECONDARY OUTCOMES:
Pain Severity | baseline, week 8, week 12, and week 24
  Pain Severity will be assessed using the 4-item Pain Severity subscale from the Brief Pain Inventory Short Form (BPI-SF). Each item is rated on a scale from 0 (no pain) to 10 (pain as bad as you can imagine), with higher scores indicating worse pain. Pain Severity will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 1 minute.
Pain Catastrophizing | baseline, week 8, week 12, and week 24
  Pain Catastrophizing will be assessed using a 13-item Pain Catastrophizing Scale (PCS) measuring the negative cognitive-emotional response to pain. Patients rate the degree to which they experience thoughts and feelings that may be associated with pain on a 0 (not at all) to 4 (all the time) scale. The PCS yields a total score and three subscales scores assessing rumination, magnification, and helplessness. It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 4 minutes.
Patient Global Impression of Change | week 8, week 12, and week 24
  Patient Global Impression of Change (PGI-C) will be assessed on a one-item scale assessing a clinically important change from the patient's perspective. Patients respond to "How would you describe your pain since you began the treatment?" on a 7-point scale ranging from "very much worse" to "very much improved." Subjects reporting "much improved" and "very much improved" will be classified as responders. The PGI-C will be administered at week 8, week 12, and week 24. Completing the survey requires approximately 1 minute.
Anxiety/Depression | baseline, week 8, week 12, and week 24
  Anxiety and Depression will be assessed on a 14-item Hospital Anxiety and Depression Scale (HADS) assessing anxiety (7 items) and depression (7 items) on a 4-point scale (0-3). Scores range from 0-21, with higher scores indicating higher symptomatology. Established cutoffs classify symptoms as not significant (0-7), subclinical (8-10), or clinically significant (11-21). The HADS will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 4 minutes.
Insomnia | baseline, week 8, week 12, and week 24
  Insomnia severity will be assessed on a 7-item Insomnia Severity Index (ISI) measuring subjective insomnia severity on a 0-4 scale, with higher scores indicating more severe insomnia symptoms. Established cutoffs classify ISI as "no clinically significant insomnia (< 8,), "subthreshold insomnia (8-14)", "clinical insomnia (moderate severity; 15-21)", and "clinical insomnia (severe, > 21)". It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 2 minutes.
Fatigue | baseline, week 8, week 12, and week 24
  Fatigue will be assessed on a 9-item Brief Fatigue Inventory (BFI) instrument assessing fatigue severity (3 items) at its "worst," "usual," and "now" during normal waking hours and amount that fatigue has interfered (6 items) with different aspects of the patient's life during the past 24 hours. Responses are measured on a 0-10 scale. Higher scores indicate worse fatigue and interference. It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 3 minutes.
Global Health | baseline, week 8, week 12, and week 24
  Global Health will be assessed using a 10-item PROMIS Global Health Scale (PROMIS-GHS) survey assessing health-related quality of life, including physical, mental, social, and overall health. Each item is rated on a 5-point scale, with higher scores indicating better overall health. It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 3 minutes.
Perceptions of aging due to arthralgia | baseline, week 8, week 12, and week 24
  Perceptions of aging due to arthralgia will be measured on a 8-item Penn Arthralgia Aging Scale (PAAS) assessing how joint pain affects body image and mental state. Each item is rated on a 0 (not at all) to 4 (completely) scale. Ratings from all items are added together to create a PAAS total score, ranging from 0 to 32. Higher scores indicate more intense perceptions of arthralgia-associated aging. It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 2 minutes.
Pleasant and painful sensations in the body | baseline, week 8, week 12, and week 24.
  Pleasant and painful sensations in the body will be measured on Sensation Manikin 2.0 (SM 2.0) - a digital, front- and back-facing human figure silhouette overlaid with a grid of 469 "sensation" pixels where patients can report the distribution of pleasant and painful sensations in the body. SM 2.0 provides three scores: 1) unpleasant sensation score representing the total body area experienced as unpleasant; 2) pleasant sensation score, representing the total body area experienced as pleasant; and 3) a sensation ratio score. It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 3 minutes.
Reappraisal | baseline, week 8, week 12, and week 24
  Reappraisal will be measured on a 9-item Mindful Reappraisal of Pain Sensations Scale (MRPS) questionnaire assessing the frequency of various forms of mindful reinterpretation of pain. Respondents rate how often they used the different ways of coping with pain in the past week on a Likert-type scale ranging from 0 (never do that) to 6 (always do that). It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 2 minutes.
Decentering | baseline, week 8, week 12, and week 24
  Decentering will be measured on a Metacognitive Processes of Decentering Scale (MPoD). The MPoD consists of the 15-item Trait (MPoD-t) and 3-item State (MPoD-s) subscales assessing decentering and the metacognitive process of decentering including meta-awareness, (dis)identification with internal experience, and (non)reactivity to internal experience. We will use the MPoD-T (Trait subscale) only. It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 2 minutes.
Nondual awareness | baseline, week 8, week 12, and week 24.
  Nondual awareness will be measured on a Nondual Awareness Dimensional Assessment (NADA) scale. The NADA consists of two measures that assess experiences of nondual awareness (NDA), including a 13-item trait-based assessment (NADA-T) and 3-item state-based assessment (NADA-S). Respondents answer each item of the NADA-T on a 5-point Likert-type scale ranging from 1 (never or very rarely) to 5 (very often or always), and each item of the NADA-S on a 11-point Likert-type scale ranging from 0 (not at all) to 10 (very much). It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 4 minutes.
Meaning in Life | baseline, week 8, week 12, and week 24
  Meaning in Life will be measured on a 10-item Meaning in Life Questionnaire (MLQ) designed to measure two dimensions of meaning in life: (1) Presence of Meaning (how much respondents feel their lives have meaning), and (2) Search for Meaning (how much respondents strive to find meaning and understanding in their lives). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (Absolutely True) to 7 (Absolutely Untrue). It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 2 minutes.
Emotion Regulation | baseline, week 8, week 12, and week 24.
  Emotion Regulation will be measured on a 10-item Emotion Regulation Questionnaire (ERQ) designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal (6 items) and (2) Expressive Suppression (4 items). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). We will use the Reappraisal subscale only (ERQ-SE). It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 2 minutes.
Savoring | baseline, week 8, week 12, and week 24
  Savoring will be measured on a 4-item Brief Savoring Inventory (BSI) scale consisting of four items that assess methods of intensifying or prolonging positive experiences by focusing on present-moment experience. Respondents answer each item on a 5-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree). It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 1 minute.
Compassion | baseline, week 8, week 12, and week 24.
  Compassion will be measured on a 5-item Compassion Subscale of Dispositional Positive Emotion Scale (CS-DPES) subscale derived from the Dispositional Positive Emotion Scale, consisting of seven subscales (joy, contentment, pride, love, compassion, amusement and awe) that measure one's dispositional tendencies to feel positive emotions towards others in their daily lives. Respondents are asked how much they identify with each of the items within each subscale (or emotions) on a 7-point Likert scale ranging from 1 (Strongly disagree) to 7 (Strongly agree). It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 1 minute.
Global self-compassion | baseline, week 8, week 12, and week 24
  Global self-compassion will be measured on a 6-item State Self-Compassion Scale (SSCS-S). Respondents answer each item of the SSCS-S on a 5-point Likert-type scale ranging from 1 (Not at all true for me) to 5 (Very true for me). It will be administered at baseline, week 8, week 12, and week 24. Completing the survey requires approximately 1 minute.
Treatment Credibility and Expectancy | baseline
  Treatment Credibility and Expectancy will be measured on a 6-item Credibility and Expectancy Questionnaire (CEQ) measuring treatment expectancy and credibility on a 9-point scale. It will be administered at baseline. Completing the survey requires approximately 1 minute.
Treatment Expectancy | baseline
  Treatment Expectancy a 4-item Treatment Expectancy Scale (TES) modified to measure MORE and SG treatment expectation. It will be administered at baseline. Completing the survey requires approximately 1 minute.
Pain Medication Diary | baseline, week 8, 12 and 24.
  Pain Medication Diaries will be administered weekly from baseline to the end of the intervention (week 8), and at weeks 12 and 24. Completing the diary requires approximately 3 minutes.
AI Adherence | baseline, week 8, 12 and 24.
  Adherence to AI will be assessed using patient EMRs, including records of treatment interruptions, premature discontinuations, and treatment changes. Self-reported adherence will be measured using the PROMIS Medication Adherence 4-item questionnaire.
Mindfulness Daily Log | weekly throughout the 8-week intervention
  The Mindfulness Daily Log tracks participants' engagement with at-home mindfulness practice, recording daily practice duration (minutes/day). This log will be collected weekly throughout the 8-week intervention for participants in the MORE treatment group. Completing the log requires approximately 1 minute.
Journaling Daily Log | weekly throughout the 8-week interventio
  The Journaling Daily Log tracks participants' engagement with at-home journaling practice, recording daily practice duration (minutes/day). This log will be collected weekly throughout the 8-week intervention for participants in the SG treatment group. Completing the log requires approximately 1 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of California San Diego (Data collection and Data analysis), San Diego, California
  - Florida State University, Tallahassee, Florida
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm